CLINICAL TRIAL: NCT01723423
Title: Mastectomy Reconstruction Outcomes Consortium (MROC) Study
Acronym: MROC
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); M.D. Anderson Cancer Center (Other); Northwestern Memorial Hospital (Other); Georgetown University (Other); Ohio State University (Other); Trinity Health Michigan (Other); Georgia Institute for Plastic Surgery (Other); Brigham and Women's Hospital (Other); University of Manitoba (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Edwin G. Wilkins, Professor of Surgery, University of Michigan
Other Study IDs: 10-PAF07150
Record Dates: First submitted 2012-02-29; First posted 2012-11-07 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; evidence based medicine; reconstruction; mastectomy; outcomes; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Expander/Implant: Patients receiving expander/implant breast reconstruction procedures.
- Lat Dorsi: Patients receiving latissimus dorsi breast reconstructions with or without implant.
- PTRAM: Patients receiving pedicle transverse rectus abdominis musculocutaneous (PTRAM)breast reconstruction.
- FTRAM: Patients receiving free transverse rectus abdominis musculocutaneous (FTRAM.)
- DIEP: Patients receiving deep inferior epigastric perforator (DIEP) breast reconstructions.
- SIEA: Patients receiving superficial inferior epigastric artery (SIEA)breast reconstruction.
- S-GAP: Patients receiving superior gluteal artery perforator breast reconstruction.
- I-GAP: Patients receiving inferior gluteal artery perforator breast reconstruction.

SUMMARY:
The MROC Study seeks to evaluate and compare from the patient's point of view the leading options for breast reconstruction after mastectomy. This study will help patients, physicians, payers and policy makers better understand the various surgeries available for breast reconstruction. Although many women choose reconstruction, the number of options as well as their pros and cons can make decision making difficult and stressful. From this research, we hope to learn more about what works best for patients undergoing these operations.

DETAILED DESCRIPTION:
Despite the growing use of breast conservation as primary therapy for breast cancer, mastectomy remains a common treatment option. Many patients choose to undergo breast reconstruction as an effective means of lessening the adverse impact of mastectomy on psychosocial functioning and quality of life. Despite these benefits, well-designed studies comparing the current choices from the patient's point of view are difficult (if not impossible) to come by. Previous research on breast reconstruction outcomes has also failed to include race and ethnicity as key variables. In order to actively participate in the reconstruction decision making process, breast cancer survivors need objective, up-to-date information on breast reconstruction outcomes from the patient's perspective.

The proposed Mastectomy Reconstruction Outcomes Consortium (MROC) Study will use a prospective cohort design to compare outcomes for the eight commonly used options for breast reconstruction: expander/implant, latissimus dorsi/implant (LD), pedicle transverse rectus abdominis musculocutaneous (PTRAM), free TRAM (FTRAM), deep inferior epigastric perforator (DIEP), superficial inferior epigastric artery (SIEA), superior gluteal artery perforator (SGAP) and inferior gluteal artery perforator (IGAP) techniques.

Outcomes assessed will include complications, postoperative pain, psychosocial well-being, physical functioning, fatigue, patient satisfaction and costs. The project will also evaluate the effects of race and ethnicity on reconstruction outcomes. Thirteen leading centers in the United States and Canada will participate. Together, these institutions perform over 3000 breast reconstructions annually. The five year study will evaluate patients preoperatively and at one week, three months, one year and two years following reconstruction. For data sources, the project will rely on medical and billing records, as well as a panel of generic and condition-specific patient-report outcome measures.

The MROC Study will benefit a variety of stakeholders in the healthcare marketplace: The project will provide consumers, providers, payers, and policy-makers with reliable, up-to-date information on the effectiveness and relative costs of surgical options for breast reconstruction, thereby promoting a more evidence-based approach to treatment and policy decision-making. Study findings will also assist health care organizations in designing systems of care tailored to the specific needs and preferences of diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Women who present themselves for reconstruction at one of 11 MROC centers
* Women undergoing one of the following types of breast reconstruction after mastectomy: tissue expander/implant, LD flap (with, or without implant), PTRAM flap, FTRAM flap, DIEP flap, S-GAP flap, I-GAP flap or SIEA flap.
* Immediate or delayed reconstruction
* Unilateral or bilateral reconstructions.
* Women receiving mastectomy for cancer prophylaxis, without history of breast cancer, will be eligible to participate.

Exclusion Criteria:

* Patients electing reconstruction following complications of breast augmentation, mastopexy (breast lift), or breast reduction will not be recruited for the study.
* Procedures performed following previously failed attempts at breast reconstruction will be excluded from the study, due to potential confounding by these previous surgeries.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing first-time breast reconstruction at one of 11 consortium sites.
Sampling Method: Non-Probability Sample
Enrollment: 4436 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health-related quality of life. | Change from baseline at 1 week, 3 months, 1 year and 2 years post-operatively.
  Patient reported outcome measures will include patient satisfaction, post-operative pain, body image, psycho-social functioning, physical functioning, and fatigue.

SECONDARY OUTCOMES:
The effects of race and ethnicity on reconstruction outcomes. | Pre-operatively and at 1 week, 3 months, 1 year and 2 years postoperatively
  Although the study will not be adequately powered to analyze outcomes by procedure type within racial and ethnic categories, we will obtain descriptive statistics for the effects of race and ethnicity on breast reconstruction outcomes.
Descriptive statistics on the relative costs of the eight procedure types. | 2 years postoperatively
  Obtain descriptive statistics on the costs of each of the seven procedure types, to gain a better understanding of the cost differences between procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin G Wilkins, MD, MS, Principal Investigator — University of Michigan; Andrea L. Pusic, MD, MHSA, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (9):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Georgia Institute for Plastic Surgery, Savannah, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - St. Joseph's Mercy Health System, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Providence Health Care - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Background] Wilkins EG, Cederna PS, Lowery JC, Davis JA, Kim HM, Roth RS, Goldfarb S, Izenberg PH, Houin HP, Shaheen KW. Prospective analysis of psychosocial outcomes in breast reconstruction: one-year postoperative results from the Michigan Breast Reconstruction Outcome Study. Plast Reconstr Surg. 2000 Oct;106(5):1014-25; discussion 1026-7. doi: 10.1097/00006534-200010000-00010. PMID 11039373
- [Background] Alderman AK, Kuhn LE, Lowery JC, Wilkins EG. Does patient satisfaction with breast reconstruction change over time? Two-year results of the Michigan Breast Reconstruction Outcomes Study. J Am Coll Surg. 2007 Jan;204(1):7-12. doi: 10.1016/j.jamcollsurg.2006.09.022. Epub 2006 Nov 16. PMID 17189107
- [Background] Alderman AK, Wilkins EG, Kim HM, Lowery JC. Complications in postmastectomy breast reconstruction: two-year results of the Michigan Breast Reconstruction Outcome Study. Plast Reconstr Surg. 2002 Jun;109(7):2265-74. doi: 10.1097/00006534-200206000-00015. PMID 12045548
- [Background] Roth RS, Lowery JC, Davis J, Wilkins EG. Persistent pain following postmastectomy breast reconstruction: long-term effects of type and timing of surgery. Ann Plast Surg. 2007 Apr;58(4):371-6. doi: 10.1097/01.sap.0000239810.38137.84. PMID 17413877
- [Background] Hu ES, Pusic AL, Waljee JF, Kuhn L, Hawley ST, Wilkins E, Alderman AK. Patient-reported aesthetic satisfaction with breast reconstruction during the long-term survivorship Period. Plast Reconstr Surg. 2009 Jul;124(1):1-8. doi: 10.1097/PRS.0b013e3181ab10b2. PMID 19568038